CLINICAL TRIAL: NCT02024724
Title: Phase 4 Study Comparing of Dexamethasone to Triamcinolone for Ultrasound-guided Trigeminal Nerve Block: A Randomized Controlled Trial.
Brief Title: Ultrasound Guided Trigeminal Nerve Block for Typical or Atypical Facial Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Antoun Nader, Professor of Anesthesiology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00083918; STU00083918 (Other: Institutional Review Board (IRB))
Record Dates: First submitted 2013-12-27; First posted 2013-12-31 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Typical Facial Pain; Atypical Facial Pain
MeSH Terms: interventions — Bupivacaine; Triamcinolone; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexamethasone (Active Comparator): 4 mg of Dexamethasone and 4 mL of 0.25% bupivacaine
  Interventions: Drug: Bupivacaine; Drug: Dexamethasone
- Triamcinolone (Active Comparator): 40 mg of Triamcinolone and 4 mL of 0.25% bupivacaine
  Interventions: Drug: Bupivacaine; Drug: Triamcinolone

INTERVENTIONS:
Drug: Bupivacaine — 4 mL of 0.25% bupivacaine
Drug: Triamcinolone — 40 mg of Triamcinolone
  Arms: Triamcinolone
Drug: Dexamethasone — 4 mg of Dexamethasone
  Arms: Dexamethasone

SUMMARY:
Trigeminal neuralgia is a craniofacial pain syndrome that is typically characterized by unilateral severe, recurrent, electrical pain in one or more distributions of the trigeminal nerve. Current treatment strategies include oral medications as first line therapy with surgical interventions reserved for those patients who are refractory to medications or unable to tolerate medication side effects. Despite these current treatment options, many patients continue to have symptoms. Ultrasound-guided trigeminal nerve block allows for fine adjustment of the needle tip and direct observation of the medicine.

Local anesthetic and steroids have been successfully used for diagnostic and or therapeutic nerve pain with great success. Steroids can be short or long acting in duration with varying side effects. If there exists a difference in duration of action, using the longer acting drug will provide a greater period of symptom relief for the patient and may allow the patient to undergo fewer interventional procedures.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to the Northwestern Pain Center who are eligible and scheduled to receive a ultrasound-guided trigeminal nerve block.

Exclusion Criteria:

* Exclusion is the same for patients who are not eligible for ultrasound guided nerve blocks.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antoun Nader, MD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Anesthesiology Pain Medcine Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2: 4 mg of Dexamethasone and 4 mL of 0.25% bupivacaine
  Bupivacaine: 4 mL of 0.25% bupivacaine
  Dexamethasone: 4 mg of Dexamethasone
- Group 1: 40 mg of Triamcinolone and 4 mL of 0.25% bupivacaine
  Bupivacaine: 4 mL of 0.25% bupivacaine
  Triamcinolone: 40 mg of Triamcinolone
Period: Overall Study
Arm/Group | Group 2 | Group 1
Started | 30 | 30
Completed | 29 | 30
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 2 | Group 1 | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 17 | 40
  >=65 years | 7 | 13 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 22 | 41
  Male | 11 | 8 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 21 | 26 | 47
  African American | 6 | 2 | 8
  Asian | 1 | 1 | 2
  Hispanic | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Subjects Reporting at Least 50% Overall Pain Relief
Description: The number of subjects reporting a minimum of 50% pain relief after receiving the injection.
Time Frame: 2 weeks
Population: Subjects reported percent relief at 2 weeks from receiving the ultrasound guided injection.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: 4 mg of Dexamethasone and 4 mL of 0.25% bupivacaine
  Bupivacaine: 4 mL of 0.25% bupivacaine
  Dexamethasone: 4 mg of Dexamethasone
- Group 2: 40 mg of Triamcinolone and 4 mL of 0.25% bupivacaine
  Bupivacaine: 4 mL of 0.25% bupivacaine
  Triamcinolone: 40 mg of Triamcinolone
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 29 | 30
Participants
  Greater than 50% Pain Relief Reported | 19 | 14
  Less than 50% Pain Relief Reported | 10 | 16
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Superiority; p = .196, Chi-squared; Median Difference (Final Values) = -30, 95% CI 2-sided [-45.00 to 10.00]

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/30
Other Adverse Events (participants affected / at risk) | 0/29 | 1/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=29) | Group 2 (N=30)
Transient numbing of the facial nerve (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes